CLINICAL TRIAL: NCT03316807
Title: Immunogenicity and Persistence of Intramuscular High Dose Recombinant Hepatitis B Vaccine in HIV-infected Adults in China
Brief Title: Immunogenicity of Hepatitis B Vaccination in HIV-infected Adults
Acronym: HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Suping Wang (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Sponsor-Investigator, Suping Wang, Professor, Shanxi Medical University
Organization: Shanxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012ZX10002001003004004
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Results first posted 2021-01-14 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-12

CONDITIONS: Hepatitis B Vaccine
Keywords: Hepatitis B, Vaccine; Randomized Controlled Trial; HIV; Immunogenicity
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60 µg dose hepatitis B vaccine (Experimental): 60 µg recombinant hepatitis B vaccine with three injections at months 0, 1, and 6
  Interventions: Biological: 60 µg dose hepatitis B vaccine
- 20 µg dose hepatitis B vaccine (Experimental): 20 µg recombinant hepatitis B vaccine with three injections at months 0, 1, and 6
  Interventions: Biological: 20 µg dose hepatitis B vaccine

INTERVENTIONS:
Biological: 60 µg dose hepatitis B vaccine — three-dose, 60 µg per dose
  Arms: 60 µg dose hepatitis B vaccine
Biological: 20 µg dose hepatitis B vaccine — three-dose, 20 µg per dose
  Arms: 20 µg dose hepatitis B vaccine

SUMMARY:
Uptake, adherence, and completion of vaccination among HIV-infected adults were low, and their immune function and immune response to hepatitis B vaccination were also suboptimal, indicating that the current practice of hepatitis B vaccination can't protect HIV-infected adults from HBV infection. And the persistence of immunity induced by hepatitis B vaccination remains a challenge.

This is a randomized, open-label trial, conducted among HIV-infected adults with drug rehabilitation. This study will compare the immunogenicity, immune persistence, and safety of three intramuscular 20µg and 60µg recombinant hepatitis B vaccines at months 0, 1, and 6 among HIV-infected adults.

DETAILED DESCRIPTION:
Participants are randomized in a ratio of 1:1 into 20 µg recombinant hepatitis B vaccine group or 60µg recombinant hepatitis B vaccine group. The 20 µg group will receive three intramuscular injections of the 20 µg recombinant hepatitis B vaccine, while the 60 µg group will receive three intramuscular injections of the 60 µg dose at months 0, 1 and 6, respectively. HBsAg and anti-HBs will be tested during the study period. Adverse reactions will be recorded after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Aged between 18 and 70 years
* Serologically negative for hepatitis B surface antigen (HBsAg) and hepatitis B surface antibody (anti-HBs) at enrollment
* Willing to adhere to the study protocol

Exclusion Criteria:

* Being pregnant
* Acute cytolysis in the last three months before enrollment
* Any vaccination before or during the month preceding enrollment
* Any Intolerance or allergy to any component of the vaccine
* Ongoing opportunistic infection
* Hematological disorder
* Cancer
* Unexplained fever the week before enrollment
* Immunosuppressive or immunomodulating treatment in the last six months
* Liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suping Wang, Principal Investigator — Shanxi Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feng Y, Yao T, Chang Y, Gao L, Shao Z, Dong S, Wu Y, Shi X, Shi J, Feng D, Cheng Y, Pan M, Li C, Wang J, Lan G, Lu H, Wang P, Xiang S, Nong L, Wang F, Liang X, Wang S. Immunogenicity and persistence of high-dose recombinant hepatitis B vaccine in adults infected with human immunodeficiency virus in China: A randomized, double-blind, parallel controlled trial. Vaccine. 2021 Jun 16;39(27):3582-3589. doi: 10.1016/j.vaccine.2021.05.044. Epub 2021 May 26. PMID 34052065

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Started | 91 | 91
Completed | 60 | 65
Not Completed | 31 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine | Total
Number analyzed (Participants) | 91 | 91 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (11.4) | 38.2 (10.6) | 39.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 33 | 75
  Male | 49 | 58 | 107
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han ethnicity | 32 | 24 | 56
  Zhuang ethnicity | 49 | 62 | 111
  others | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Anti-HBs Seroconversion at Month 7
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA(Chemiluminescent Microparticle Immunoassay ). The accepted protective serum anti-HBs level was ≥10 mIU/ml.
Time Frame: Month 7
Population: 83 and 82 patients in the IM60（60μg recombinant hepatitis B vaccine） and IM20（20μg recombinant hepatitis B vaccine） groups completed the followed-up at months 7.
Measure: Count of Participants; unit: Participants
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 83 | 82
Participants | 75 | 69

2. Secondary Outcome: Anti-HBs Concentration at Month 7
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA(Chemiluminescent Microparticle Immunoassay ).
Time Frame: Month 7
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 83 | 82
mIU/mL | 623.3 [427.7 to 836.9] | 469.4 [326.8 to 611.9]

3. Secondary Outcome: Number and Percentage of Participants With Anti-HBs Seroconversion at Month 12
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA（Chemiluminescent Microparticle Immunoassay）.The accepted protective serum anti-HBs level was ≥10 mIU/ml.
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 74 | 68
Participants | 55 | 50

4. Secondary Outcome: Anti-HBs Concentration at Month 12
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA（Chemiluminescent Microparticle Immunoassay）.
Time Frame: Month 12
Measure: Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 74 | 68
mIU/ml | 290.4 [132.6 to 448.1] | 264.4 [95.3 to 433.4]

5. Secondary Outcome: Occurrence of Adverse Events After Vaccination
Description: Occurrence of adverse reactions within 7 days after vaccination with the hepatitis B vaccine
Time Frame: Within 7 days after the vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 88 | 88
Participants
  pain | 5 | 5
  erythema | 6 | 5
  edema | 5 | 4
  induration | 4 | 4

6. Secondary Outcome: Occurrence of Adverse Events After Vaccination
Description: Occurrence of adverse reactions within 28 days after vaccination with the hepatitis B vaccine
Time Frame: Within 28 days after vaccination
Population: Safety analysis was performed on all included participants.
Measure: Number; unit: participants
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 88 | 88
participants
  fever | 1 | 1
  headache | 2 | 1

7. Secondary Outcome: Serious Adverse Events (SAE) Occurred During 42 Month
Description: Occurrence of Serious adverse events (SAE) within 42 month after vaccination with the hepatitis B
Time Frame: Month 0-42
Measure: Count of Participants; unit: Participants
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 88 | 88
Participants | 0 | 0

8. Other Pre Specified Outcome: Number and Percentage of Participants With Anti-HBs High-level Response at Month 7
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA. and anti-HBs concentrations ≥100 mIU/ml were high-level response.
Time Frame: Month 7
Measure: Count of Participants; unit: Participants
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 83 | 82
Participants | 62 | 54

9. Other Pre Specified Outcome: Number and Percentage of Participants With Anti-HBs High-level Response at Month 12
Description: as for outcome 8
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 74 | 68
Participants | 34 | 26

10. Other Pre Specified Outcome: Number and Percentage of Participants With Anti-HBs Antibodies at Month 6 Before the Third Injection
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA. The accepted protective serum anti-HBs level was ≥10 mIU/ml.
Time Frame: Month 6 before the third injection
Population: 83 and 70 patients in the IM60 and IM20 groups completed the followed-up at month 6 before the third injection.
Measure: Count of Participants; unit: Participants
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 83 | 80
Participants | 65 | 61

11. Other Pre Specified Outcome: Anti-HBs Concentration at Month 6 Before the Third Injection
Description: Anti-HBs concentration at month 6 before the third injection as measured by CMIA（Chemiluminescent Microparticle Immunoassay）.
Time Frame: Month 6 before the third injection
Measure: Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 83 | 80
mIU/ml | 148.9 [78.1 to 219.7] | 130.6 [72.5 to 188.8]

12. Other Pre Specified Outcome: Number and Percentage of Participants With Anti-HBs High-level Response at Month 6 Before the Third Injection
Description: as for outcome 8
Time Frame: Month 6 before the third injection
Measure: Count of Participants; unit: Participants
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 83 | 80
Participants | 29 | 27

13. Other Pre Specified Outcome: Number and Percentage of Participants With Anti-HBs Seroconversion at Month 42
Description: as for outcome 1
Time Frame: Month 42
Measure: Count of Participants; unit: Participants
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
Number analyzed (Participants) | 60 | 65
Participants | 31 | 29

ADVERSE EVENTS:
Arm/Group | 60 µg Dose Hepatitis B Vaccine | 20 µg Dose Hepatitis B Vaccine
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/88
Other Adverse Events (participants affected / at risk) | 8/88 | 6/88
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 60 µg Dose Hepatitis B Vaccine (N=88) | 20 µg Dose Hepatitis B Vaccine (N=88)
Pain (Musculoskeletal and connective tissue disorders) | 5 | 5
erythema (Skin and subcutaneous tissue disorders) | 6 | 5
edema (Skin and subcutaneous tissue disorders) | 5 | 4
induration (Skin and subcutaneous tissue disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No